CLINICAL TRIAL: NCT06498713
Title: Patient Controlled Self-Administration of Oral Liquid Medication: Acetaminophen Trial
Brief Title: Patient Controlled Administration of Liquid Acetaminophen
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000037919
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Pain; Pain, Postoperative
Keywords: Pain Management
MeSH Terms: conditions — Pain; Pain, Postoperative; Agnosia | interventions — Acetaminophen; Tablets; Fluid Therapy

STUDY DESIGN:
Intervention Model Description: Patients undergoing total shoulder arthroplasty or reverse total shoulder arthroplasty at Yale New Haven Hospital at St. Raphael's Campus.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Nurse Administered Acetaminophen (Active Comparator): Participants will receive acetaminophen pills 650 mg every 4 hours as needed (PRN) administered by nurse per standard of care
  Interventions: Drug: Acetaminophen 650 mg Oral Tablet
- CADD pump Administered Acetaminophen (Participant Controlled) (Experimental): Participants will receive a CADD pump primed and programmed to deliver 650 mg liquid acetaminophen into a medication cup every 4 hours as needed (PRN).
  Interventions: Drug: Acetaminophen 650mg Liquid; Device: CADD pump

INTERVENTIONS:
Drug: Acetaminophen 650 mg Oral Tablet — 650 mg pills
  Other Names: Tylenol
  Arms: Nurse Administered Acetaminophen
Drug: Acetaminophen 650mg Liquid — 650 mg liquid
  Other Names: Tylenol
  Arms: CADD pump Administered Acetaminophen (Participant Controlled)
Device: CADD pump — Primed and programmed to delivery 650 mg liquid acetaminophen into a medication cup every 4 hours as needed.
  Arms: CADD pump Administered Acetaminophen (Participant Controlled)

SUMMARY:
This is a proof of concept pilot study investigating the feasibility and acceptability of patient controlled oral medication administration, using the commonly used and low risk medication in the hospital, oral acetaminophen.

DETAILED DESCRIPTION:
The primary objective of this prospective pilot study is to determine the feasibility of patient-controlled administration of liquid oral acetaminophen using recruitment rate and adherence to the study protocol rate as surrogate markers. Investigators hypothesize that patients will accept the new concept of self-controlled oral administration of liquid acetaminophen, with more than 50% patient enrollment rate and less than 20% withdrawal rate from the study group to the traditional nurse-administered acetaminophen pills.

The secondary objective of this study is to determine the preliminary efficacy of patient-controlled delivery of oral acetaminophen administration.

If the medication is spilled or otherwise not dispensed correctly, the patients will be instructed to report this instantly to the nurse. The nurse will document and provide a replacement.

All study participants have the option to call the nurse for assistance with break through pain. In addition, there is a call button to call for help with any other needs or discomfort.

All other medications, such as NSAIDs or oral opioids, will be administered as prescribed.

Participants will have to fill out a paper questionnaire and keep a pain diary, and nurses will have to fill out a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Participants

* Adult patients older than 18 years old admitted to SRC for total shoulder and reverse total shoulder arthroplasty

Nurses

* The nurse who will administer acetaminophen to a study patient.

Exclusion Criteria:

Participants

* Pregnant patient
* Patients that cannot swallow pills or cannot take liquid (for example due to risk of aspiration)
* Emergency surgery
* Chronic pain
* On home opioids, any other pain modulating medications including benzodiazepine, Neurontin, ketamine.
* Past medical or social history of substance abuse disorder, including ethanol misuse disorder, marijuana misuse disorder
* History of any psychiatric disorders including anxiety, depression, any cognitive dysfunction
* Any patients who cannot provide informed consents on their own (those who would need Legally Authorized Representatives (LARs) or surrogates)
* Liver dysfunction limiting amount of safe oral acetaminophen
* baseline hyperbilirubinemia (ex: chronic liver disease, Gilbert's)
* patients unable to take PO
* Patients with neurologic, neuromuscular, or movement disorders unable to drink from a cup.

Nurses

* any nurse who is not involved in the direct care of a study patient, or who is not comfortable with setting up the PCA pump.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Participant enrollment rate | up to 12 months
  The percentage of participants that enroll
Participant adherence to the study protocol | up to 12 months
  Percentage of participants that withdraw from treatment group, i.e. switch from patient controlled liquid group to the nurse-administered pill control group
Nurse Questionnaire | Study day 0, 1, 2 and 3
  Nurse ranking of patient controlled liquid oral acetaminophen vs. nurse-administered pill acetaminophen. (Mean score, Total Scale of 0-10: 0: much worse; 5:same; 10: much better)

SECONDARY OUTCOMES:
Mean daily acetaminophen consumption | 12 months
  Mean daily acetaminophen consumption in milligrams collected using the electronic medical record
Mean Pain score | 12 months
  Participants will be asked via Pain Diary to rate their pain using numeric pain scores from 0 to 10, 0 as no pain, 10 is the worst possible.
Mean time to medication delivery | 12 months
  Medication delivery: Mean time in minutes from the time when pain medication requested by the participant to the time pain medication is delivered

CONTACTS AND LOCATIONS:
Overall Officials: Jinlei Li, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital at St. Raphael's Campus, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No